CLINICAL TRIAL: NCT02148380
Title: Combination of Chemotherapy and Gefitinib as First-line Treatment of Patients With Advanced Lung Adenocarcinoma and Sensitive EGFR Mutations: a Randomised Controlled Trial
Brief Title: Combination of Chemotherapy and Gefitinib as First-line Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baohui Han (Other)
Responsible Party: Sponsor-Investigator, Baohui Han, the chief physician, Shanghai Chest Hospital
Organization: Shanghai Chest Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: chest20140001
Record Dates: First submitted 2014-05-21; First posted 2014-05-28 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Non-Small-Cell Lung Cancer
Keywords: Lung adenocarcinoma,EGFR mutation, chemotherapy, gefitinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Carboplatin; Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- chemotherapy group(B) (Experimental): pemetrexed plus carboplatin pemetrexed (500 mg/m(2) on day 1) plus carboplatin (AUC 5 on day 1) every 4 weeks for up to six cycles, then continued to receive pemetrexed(500 mg/m(2) on day 1) alone every 4 weeks
  Interventions: Drug: pemetrexed plus carboplatin
- combination therapy group(A) (Experimental): pemetrexed (500 mg/m(2) on day 1) plus carboplatin (AUC 5 on day 1) combined with gefitinib (250 mg/day on days 5-21) and repeated every 4 weeks for up to six cycles,then continued to receive pemetrexed combined with gefitinib every 4 weeks.
  Interventions: Drug: pemetrexed plus carboplatin; Drug: gefitinib
- gefitinib group (group C) (Experimental): received gefitinib( 250 mg/day)alone. All therapies of 3 groups were continued until progression or unacceptable toxicity or death
  Interventions: Drug: gefitinib

INTERVENTIONS:
Drug: pemetrexed plus carboplatin
  Other Names: Alimita plus carboplatin
  Arms: chemotherapy group(B); combination therapy group(A)
Drug: gefitinib
  Other Names: Iressa
  Arms: combination therapy group(A); gefitinib group (group C)

SUMMARY:
The results of fastact2 show that chemotherapy plus erlotinib significantly prolonged PFS and OS of patients with NSCLC. However, outcome of the combination therapy are similar to those reported in several trials of single-agent EGFR TKIs. So which is the optimal first-line treatment for patients who harbored a sensitive EGFR mutation? The investigators need a head-to-head study to reply.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Age >=18 years
3. Histologically documented, unresectable, inoperable, locally advanced, recurrent or metastatic Stage IV Non-Small Cell Lung Cancer (NSCLC)
4. A cytologic diagnosis is acceptable (i.e., FNA or pleural fluid cytology)
5. Measurable or non-measurable disease
6. Able to comply with study and follow-up procedures

Exclusion Criteria:

* Evidence of small cell, carcinoid, or mixed small cell/non-small cell histology
* Malignancies within 3 years except for adequately treated carcinoma in situ of -the cervix or basal or squamous cell skin cancer
* Symptomatic or untreated brain metastases
* Prior systemic chemotherapy for NSCLC
* Unstable systemic disease, including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, or myocardial infarction within 6 months prior to Day 1, or serious cardiac arrhythmia requiring medication (patients with chronic atrial arrhythmia, i.e., atrial fibrillation or paroxysmal supraventricular tachycardia, are eligible)
* History of other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect the interpretation of the results of the study or render the patient at high risk from treatment complications
* Gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for intravenous (IV) alimentation, or prior surgical procedures affecting absorption
* Pregnancy or lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2014-05; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
progression-free survival | 6-month

SECONDARY OUTCOMES:
overall survival | 2 years
to evaluate the safety profile between three groups | 6 months
  Toxicity will be graded according to NCI CTCAE, version 4.0. The analysis of safety/tolerability data will be descriptive; toxicity events will be individually tabulated.

CONTACTS AND LOCATIONS:
Overall Officials: Baohui Han, Dr, Study Chair — Vice President of Shanghai Chest Hospital,Sponsor of study; Bo Jin, Dr, Study Director — Study Leader,Doctor of Shanghai Chest Hospital; Yanjie Niu, Master, Principal Investigator — Doctor of Shanghai Chest Hospital; Yanwei Zhang, Dr, Principal Investigator — Doctor of Shanghai Chest Hospital; Tianqing Chu, Dr, Principal Investigator — Doctor of Shanghai Chest Hospital; Aiqin Gu, Master, Principal Investigator — Doctor of Shanghai Chest Hospital; Lei Zhu, Master, Principal Investigator — Doctor of Shanghai Chest Hospital; Jun Pei, Principal Investigator — Doctor of Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lou Y, Xu J, Zhang Y, Lu J, Chu T, Zhang X, Wang H, Zhong H, Zhang W, Han B. Chemotherapy Plus EGFR-TKI as First-Line Treatment Provides Better Survival for Advanced EGFR-Positive Lung Adenocarcinoma Patients: Updated Data and Exploratory In Vitro Study. Target Oncol. 2020 Apr;15(2):175-184. doi: 10.1007/s11523-020-00708-y. PMID 32170554